CLINICAL TRIAL: NCT06855836
Title: Efficacy and Implementation Considerations for a Peer-led Motivational Interviewing Intervention to Promote Uptake of Drug Checking Services and Safe Drug Use Behaviors to Reduce Overdose
Brief Title: Motivational Interviewing to Increase Uptake of Drug Checking and Safe Drug Use Behaviors to Reduce Overdose
Acronym: MI-CHANCE
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Diego (Other)
Collaborators: Harm Reduction Coalition of San Diego (HRCSD) (Unknown)
Responsible Party: Principal Investigator, Steffanie Strathdee, Harold Simon Distinguished Professor, Co-director, Center for Innovative Phage Applications & Therapeutics (IPATH) Division of Infectious Diseases and Global Public Health Department of Medicine, UC San Diego Health Sciences, University of California, San Diego
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 1R33DA061260-01 (NIH)
Record Dates: First submitted 2025-02-25; First posted 2025-03-04 (Actual); Last update posted 2025-12-12 (Actual); Status verified 2025-12

CONDITIONS: Overdose
MeSH Terms: conditions — Drug Overdose | interventions — Spectroscopy, Fourier Transform Infrared; Motivational Interviewing; Influenza Vaccines

STUDY DESIGN:
Intervention Model Description: All recruited study participants will receive the Overdose Education and Naloxone Distribution (OEND) materials. The control group will receive additional Flu and Hepatitis A education as Group 1, and the experimental group will receive the MI-CHANCE intervention as Group 2
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard of Care Control (SOC; Group 1) -TS + FTIR + Flu and Hepatitis A education. (Placebo Comparator): Participants will receive naloxone, overdose prevention pamphlets and be shown videos (English or Spanish) on how naloxone works. Participants will be offered the services of drug sample testing by CheckSD's technician after their study session. The training videos will be on Flu and Hepatitis A education. Overall, the session for Group 1 as the attention control participants will last 30 minutes.
  Interventions: Behavioral: TS + FTIR + Flu and Hepatitis A Education
- MI-CHANCE Intervention (Group 2) - TS+FTIR+MI. (Experimental): Participants will receive naloxone, overdose prevention pamphlets and MI in a 30-minute counseling session. Trained peer-support specialists will engage participants in discussion on the drug supply, ask to rate how certain they are about their drugs' content, how they perceive their OD risk, and shown a brief video about FTIR. Using "decisional balance", participants will identify pros and cons of regularly using DCS prior to drug use and modifying drug use behaviors based on their own potential safer alternatives. Once the balance shifts towards positive change, they will be offered to get their own drug tested by CheckSD's technician and provided with results highlighting drug potency and purity. If they decline, a dummy sample containing fentanyl will be used. Participants will develop an action plan with harm reduction principles to problem-solve specific challenges, identify their goals to use DCS and prevent OD.
  Interventions: Behavioral: MI-CHANCE (TS + FTIR + MI)

INTERVENTIONS:
Behavioral: MI-CHANCE (TS + FTIR + MI) — MI-CHANCE was built following key principles of MI (partnership, acceptance, compassion and evocation) to empower PWUD, help them identify potential benefits of DCS and strategies to integrate these into their daily lives. The manual follows three key stages: 1) introducing DCS, 2) generating change talk, and 3) verbalizing commitment, using open questions, affirmations, reflections and summaries. Pros and cons for regularly using CheckSD and changing drug use behaviors accordingly were identified in the literature and through discussions with PWUD and HRCSD staff. Peer support specialists are urged to mirror participants' own language (e.g., oxy or M30s=oxycontin; carga= heroin; malilla=withdrawal, fetty=fentanyl). Challenges were categorized into 8 key areas: legal, financial, scheduling, transportation, ability to change drug use behaviors, communication with SSP staff, managing mood and substance use.
  Other Names: Motivational Interviewing
  Arms: MI-CHANCE Intervention (Group 2) - TS+FTIR+MI.
Behavioral: TS + FTIR + Flu and Hepatitis A Education — Naloxone and educational materials (i.e. pamphlets) on overdose prevention, videos (English or Spanish) on naloxone, flu and Hepatitis A education.
  Arms: Standard of Care Control (SOC; Group 1) -TS + FTIR + Flu and Hepatitis A education.

SUMMARY:
A hybrid type 1 study will be conducted to evaluate efficacy and preliminary implementation considerations for a novel intervention to promote uptake of drug checking services (DCS) and safer drug use behaviors among people who use drugs (PWUD) to reduce incidence of overdose (OD) and HIV and Hepatitis C virus (HCV) infections in San Diego County.

Along with ~50 other syringe services programs (SSPs) in the US, the Harm Reduction Coalition San Diego (HRCSD), a local SSP, recently launched CheckSD (San Diego), a DCS using test strips (TS) and Fourier Transform Infrared Spectrometry (FTIR) that allows people to submit drug samples with non-nominal identifiers and obtain personalized results. While most existing DCS using FTIR offer some counseling, no theory-based interventions to increase DCS uptake and promote post-DCS adoption of safer drug use behaviors have been rigorously evaluated

DETAILED DESCRIPTION:
588 PWUD who have not yet used CheckSD will be recruited into a two-arm randomized controlled trial (RCT) (N=294 per group). Recruitment sources will be the community and La Frontera study. Both arms will have access to CheckSD's standard of care (SOC) already available at SSP sites (i.e., FTIR, and overdose education and naloxone distribution (OEND)). PWUD randomized to receive MI-CHANCE will receive it from HRCSD's peer counselors who will be trained in motivational interviewing (MI) to encourage CheckSD uptake and safer drug use behaviors. Those in the attention-control SOC arm will receive Flu and Hepatitis A education. All will undergo semi-annual follow-up for 30 months.

Primary Objective: To test the efficacy of MI-CHANCE on reducing rates of combined fatal and non-fatal OD over 30 months and examine social cognitive theory (SCT)-informed mediators and moderators of intervention effects (i.e., knowledge, outcome expectancies, self-efficacy)

ELIGIBILITY:
Inclusion Criteria:

A total of 588 PWUD participants will be recruited for the proposed study (MI-CHANCE). To be eligible to participate in this study, an individual must meet all of the following criteria:

1. Provision of signed and dated informed consent form
2. Stated willingness to comply with all study procedures and availability for the duration of the study
3. Be aged ≥18 years at time of recruitment
4. Must have used illicit opiates (e.g., heroin, fentanyl) and/or methamphetamine ≤1 week prior to recruitment date
5. Live in San Diego County with no plans to permanently move over the next 30 months
6. Have not previously used the CheckSD drug checking service
7. Enrolled into ongoing prospective cohort study La Frontera (the border) (existing or new participants)

Enrollment will be capped so that <25% of the sample reports only using methamphetamine to ensure that the sample is comprised primarily of people who use opiates who are at greatest risk of OD. Recruitment will be done through targeted sampling at hotspots as well as homeless encampments, shelters and outreach through social media.

Exclusion Criteria:

An individual who meets any of the following criteria will be excluded from participation in this study:

1. Not being able to provide a signed and dated informed consent form
2. Not willing to comply with all study procedures and availability for the duration of the study
3. Currently enrolled in another randomized controlled trial
4. Not having used illicit opiates (e.g., heroin, fentanyl), methamphetamine ≤1 week prior to recruitment date
5. Having used CheckSD (i.e. drug testing with TS+FTIR)
6. Participated in the MI-CHANCE pilot

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 588 (Actual)
Dates: Start 2025-03-03 (Actual); Primary Completion 2029-02 (Estimated); Study Completion 2029-05 (Estimated)

PRIMARY OUTCOMES:
Risk rates of fatal and non-fatal overdose over 30 months | Through study completion, an average of 30 months
  Rate of fatal and non-fatal ODs over the course of the study (i.e., the total # of ODs that a participant experiences during the study offset by the natural log of the time spent at risk during the study). Self-reported and obtained through record linkage between MI-CHANCE and emergency medical services and the medical examiner's office to obtain data on ODs that received medical attention and OD deaths, respectively

SECONDARY OUTCOMES:
Frequency of drug checking service utilization | At baseline and every 6 months for 30 months
  Number of times one utilized CheckSD over the past 6 months. Self-reported
Risk rates of HIV/HCV infection over 30 months | Through study completion, an average of 30 months
  Rates of HIV and HCV infection determined through serology (biological sample collection) over the course of the study (i.e. between baseline and 30 months)

CONTACTS AND LOCATIONS:
Locations (1):
- MI CHANCE - Park Blvd, San Diego, California, United States

REFERENCES:
- [Background] Geldhof, G. J., Anthony, K. P., Selig, J. P., & Mendez-Luck, C. A. (2018). Accommodating binary and count variables in mediation: A case for conditional indirect effects. International Journal of Behavioral Development, 42(2), 300-308. https://doi.org/10.1177/0165025417727876
- [Background] Friedman J, Godvin M, Molina C, Romero R, Borquez A, Avra T, Goodman-Meza D, Strathdee S, Bourgois P, Shover CL. Fentanyl, heroin, and methamphetamine-based counterfeit pills sold at tourist-oriented pharmacies in Mexico: An ethnographic and drug checking study. Drug Alcohol Depend. 2023 Aug 1;249:110819. doi: 10.1016/j.drugalcdep.2023.110819. Epub 2023 Jun 9. PMID 37348270
- [Background] Alexander RS, Canver BR, Sue KL, Morford KL. Xylazine and Overdoses: Trends, Concerns, and Recommendations. Am J Public Health. 2022 Aug;112(8):1212-1216. doi: 10.2105/AJPH.2022.306881. PMID 35830662
- [Background] Friedman J, Montero F, Bourgois P, Wahbi R, Dye D, Goodman-Meza D, Shover C. Xylazine spreads across the US: A growing component of the increasingly synthetic and polysubstance overdose crisis. Drug Alcohol Depend. 2022 Apr 1;233:109380. doi: 10.1016/j.drugalcdep.2022.109380. Epub 2022 Feb 26. PMID 35247724
- [Background] Roberts A, Korona-Bailey J, Mukhopadhyay S. Notes from the Field: Nitazene-Related Deaths - Tennessee, 2019-2021. MMWR Morb Mortal Wkly Rep. 2022 Sep 16;71(37):1196-1197. doi: 10.15585/mmwr.mm7137a5. No abstract available. PMID 36107790
- [Background] Riggins A. Dangerous mix of fentanyl and animal tranquilizer detected in few seizures in San Diego. San Diego Union Tribune, January 16, 2023
- [Background] Riggins A. San Diego man sentenced in fentanyl-xylazine case as local evidence of dangerous 'tranq' drug grows. San Diego Union Tribune, September 9, 2023.
- [Background] Volkow ND, Califf RM, Sokolowska M, Tabak LA, Compton WM. Testing for Fentanyl - Urgent Need for Practice-Relevant and Public Health Research. N Engl J Med. 2023 Jun 15;388(24):2214-2217. doi: 10.1056/NEJMp2302857. Epub 2023 Jun 10. No abstract available. PMID 37306505
- [Background] California Health and Safety Code. Division 10. Uniform controlled substances act [11000 - 11651]. Chapter 6. Offenses and penalties [11350 - 11392] Article 4. Miscellaneous Offenses and Provisions [11364 - 11376.5]. 1972.
- [Background] California Health and Safety Code. Division 105. Communicable disease prevention and control [120100 - 122420]. Part 4. Human immunodeficiency virus (HIV) [120775 - 121349.3]. Chapter 18. Clean Needle and Syringe Exchange Program [121349 - 121349.3]. 1972.
- [Background] Davis CS, Lieberman AJ, O'Kelley-Bangsberg M. Legality of drug checking equipment in the United States: A systematic legal analysis. Drug Alcohol Depend. 2022 May 1;234:109425. doi: 10.1016/j.drugalcdep.2022.109425. Epub 2022 Mar 22. PMID 35344879
- [Background] Controlled substances: paraphernalia: controlled substance testing.; 2022. https://leginfo.legislature.ca.gov/faces/billNavClient.xhtml?bill_id=202120220AB1598.
- [Background] Green TC, Park JN, Gilbert M, McKenzie M, Struth E, Lucas R, Clarke W, Sherman SG. An assessment of the limits of detection, sensitivity and specificity of three devices for public health-based drug checking of fentanyl in street-acquired samples. Int J Drug Policy. 2020 Mar;77:102661. doi: 10.1016/j.drugpo.2020.102661. Epub 2020 Jan 14. PMID 31951925
- [Background] McCrae K, Tobias S, Grant C, Lysyshyn M, Laing R, Wood E, Ti L. Assessing the limit of detection of Fourier-transform infrared spectroscopy and immunoassay strips for fentanyl in a real-world setting. Drug Alcohol Rev. 2020 Jan;39(1):98-102. doi: 10.1111/dar.13004. Epub 2019 Nov 19. PMID 31746056
- [Background] Ti L, Tobias S, Lysyshyn M, Laing R, Nosova E, Choi J, Arredondo J, McCrae K, Tupper K, Wood E. Detecting fentanyl using point-of-care drug checking technologies: A validation study. Drug Alcohol Depend. 2020 Jul 1;212:108006. doi: 10.1016/j.drugalcdep.2020.108006. Epub 2020 May 12. PMID 32438280
- [Background] Tupper KW, McCrae K, Garber I, Lysyshyn M, Wood E. Initial results of a drug checking pilot program to detect fentanyl adulteration in a Canadian setting. Drug Alcohol Depend. 2018 Sep 1;190:242-245. doi: 10.1016/j.drugalcdep.2018.06.020. Epub 2018 Jul 24. PMID 30064061
- [Background] Carroll JJ, Mackin S, Schmidt C, McKenzie M, Green TC. The Bronze Age of drug checking: barriers and facilitators to implementing advanced drug checking amidst police violence and COVID-19. Harm Reduct J. 2022 Feb 4;19(1):9. doi: 10.1186/s12954-022-00590-z. PMID 35120531
- [Background] Wallace B, van Roode T, Pagan F, Phillips P, Wagner H, Calder S, Aasen J, Pauly B, Hore D. What is needed for implementing drug checking services in the context of the overdose crisis? A qualitative study to explore perspectives of potential service users. Harm Reduct J. 2020 May 12;17(1):29. doi: 10.1186/s12954-020-00373-4. PMID 32398090
- [Background] Glick JL, Christensen T, Park JN, McKenzie M, Green TC, Sherman SG. Stakeholder perspectives on implementing fentanyl drug checking: Results from a multi-site study. Drug Alcohol Depend. 2019 Jan 1;194:527-532. doi: 10.1016/j.drugalcdep.2018.10.017. Epub 2018 Nov 13. PMID 30551090
- [Background] Administration SAaMHS. The Opioid Crisis and the Hispanic/Latino Population: An Urgent Issue, 2020
- [Background] Rosales R, Janssen T, Yermash J, Yap KR, Ball EL, Hartzler B, Garner BR, Becker SJ. Persons from racial and ethnic minority groups receiving medication for opioid use disorder experienced increased difficulty accessing harm reduction services during COVID-19. J Subst Abuse Treat. 2022 Jan;132:108648. doi: 10.1016/j.jsat.2021.108648. Epub 2021 Oct 30. PMID 34742607
- [Background] Friedman JR, Hansen H. Evaluation of Increases in Drug Overdose Mortality Rates in the US by Race and Ethnicity Before and During the COVID-19 Pandemic. JAMA Psychiatry. 2022 Apr 1;79(4):379-381. doi: 10.1001/jamapsychiatry.2022.0004. PMID 35234815
- [Background] Kaiser Family Foundation. Opioid Overdose Deaths by Race/Ethnicity. https://www.kff.org/other/stateindicator/
- [Derived] Bailey K, Strathdee SA, Bazzi AR, Stamos-Buesig T, Godvin M, Harvey-Vera A, Abramovitz D, Vera CF, Patterson TL, Davidson PJ, Borquez A. Motivational interviewing to increase drug checking and reduce overdose rates among people who use drugs: protocol for a hybrid type 1 effectiveness-implementation trial of an adjunctive intervention. BMC Public Health. 2025 Sep 30;25(1):3228. doi: 10.1186/s12889-025-24460-y. PMID 41029610

DOCUMENTS (1):
  • Informed Consent Form (2025-05-13): https://cdn.clinicaltrials.gov/large-docs/36/NCT06855836/ICF_000.pdf